CLINICAL TRIAL: NCT06810076
Title: Developing and Evaluating a Machine-Learning Opioid Prediction & Risk-Stratification E-Platform (DEMONSTRATE)
Brief Title: Developing and Evaluating a Machine-Learning Opioid Overdose Prediction & Risk-Stratification Tool in Primary Care
Acronym: DEMONSTRATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Applied Decision Science (Unknown)
Responsible Party: Principal Investigator, Wei-Hsuan Lo-Ciganic, Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY24040038; R01DA050676 (NIH)
Record Dates: First submitted 2025-01-27; First posted 2025-02-05 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Opiate Overdose; Opioid-Related Disorders; Narcotic-Related Disorders; Substance-related Disorders; Chemically-Induced Disorders; Mental Disorders
Keywords: Opiate overdose; Opioid-Related Disorders; Risk Evaluation and Mitigation; Machine Learning; Medical Order Entry Systems; Decision Support Systems, Clinical
MeSH Terms: conditions — Opiate Overdose; Opioid-Related Disorders; Narcotic-Related Disorders; Substance-Related Disorders; Chemically-Induced Disorders; Mental Disorders | interventions — Methods

STUDY DESIGN:
Intervention Model Description: This single-arm clinical trial employs a pre- and post-implementation pilot evaluation design to assess the usability, acceptability, and feasibility of implementing a ML-driven overdose CDS tool across thirteen UF Health primary care clinics (3 internal medicine and 6 family medicine clinics in Gainesville, Florida). The CDS tool will generate an Overdose Prevention Alert (OPA) when a PCP signs an opioid order in Epic® for patients at elevated risk of opioid overdose identified by ML algorithm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Overdose Prevention Alert (OPA) Intervention Arm (Experimental): The intervention arm will receive a ML CDS tool that provides interruptive alerts for patients at elevated risk of opioid overdose, triggered when a clinician signs an opioid order.
  Interventions: Behavioral: Machine Learning-Based Clinical Decision Support: Overdose Prevention Alert (OPA) Intervention

INTERVENTIONS:
Behavioral: Machine Learning-Based Clinical Decision Support: Overdose Prevention Alert (OPA) Intervention — In this study, researchers will pilot test an interruptive, ML CDS tool for opioid overdose risk across thirteen primary care clinics at the UF Health in Gainesville, FL. When a patient is identified by the ML algorithm as having an elevated overdose risk and a PCP signs an opioid prescription for the patient, an Opioid Prevention Alert (OPA) will be triggered. The alert will include the rationale for the patient's elevated risk status and provide three risk mitigation recommendations: optimizing pain treatment and mental health support, reviewing and discussing risks with the patient, and offering naloxone annually if no prior naloxone order is found in the patient's record. PCPs can also select an override reason, such as the patient already has naloxone, declined the intervention, is not present/it is not the right time, or the alert is not relevant/other comments, when appropriate.

SUMMARY:
This clinical trial aims to evaluate the pilot implementation of a machine-learning (ML)-driven clinical decision support (CDS) tool designed to predict opioid overdose risk within the electronic health record (EHR) system at UF Health Internal Medicine and Family Medicine clinics in Gainesville, Florida. The study will use a pre- versus post-implementation design to compare outcomes within clinics, focusing on measures such as naloxone prescribing rates and opioid overdose occurrences. Researchers will also assess the usability, acceptability, and feasibility of the CDS tool through qualitative interviews with primary care clinicians (PCPs) in the participating clinics.

DETAILED DESCRIPTION:
This clinical trial evaluates the pilot implementation of a ML-driven CDS tool designed to predict opioid overdose risk within the electronic health record (EHR) system at thirteen UF Health internal medicine and family medicine clinics in Gainesville, Florida.

The implementation process involved backend and frontend development and integration of the CDS tool. For backend integration, the investigators reviewed clinical workflows, designed a data flow plan to incorporate risk scores into patient charts, and collaborated with UF Health IT and Integrated Data Repository (IDR) Research Services to address alert implementation, data flow, server specifications, and responsibilities. Risk assessments approved by UF Health IT and the institutional review board (IRB) ensured secure access to patient health information (PHI) and enabled EHR integration. For frontend development, the investigators used a user-centered design approach to create the CDS tool prototype, incorporating feedback from PCPs during formative interviews to refine the user interface and ensure timely, actionable alerts through the EPIC system without disrupting clinical workflows.

The study primarily aims to assess the usability, acceptance, and feasibility of the CDS tool six months post-implementation through mixed-method evaluations. Researchers will use semi-structured interviews and an online questionnaire to collect feedback from PCPs, focusing on alert usability, preferences, and outcomes. Quantitative analyses will evaluate alert penetration, usage patterns, and PCP actions, while qualitative analyses will explore themes and insights from override comments to guide tool optimization. Researchers will also explore secondary patient-level outcomes using EHR data such as naloxone prescriptions.

ELIGIBILITY:
Inclusion Criteria:

For PCP level outcomes assessment

* PCPs
* practicing in any of the 13 participating clinics (10 UF Health Family Medicine clinics and 3 UF Health Internal Medicine) in Gainesville, Florida.

For patient level outcomes assessment:

Inclusion criteria: Patients who seen in any of the 9 participating UF Health clinics who

* are aged ≥18 years
* received any opioid prescription in the past year prior to their clinic visit.
* are identified as being at elevated risk for overdose by the ML algorithm. Exclusion Criteria: Patients who
* had malignant cancer diagnosis or hospice care prior to study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2026-04-07 (Estimated); Study Completion 2026-10-02 (Estimated)

PRIMARY OUTCOMES:
Composite patient-level outcomes related to opioids | From enrollment and up to 12 months (3, 6, 12 months) post implementation of the OPA
  The CDS tool will generate an Overdose Prevention Alert (OPA) when a PCP signs an opioid order in Epic®. To evaluate the tool's effectiveness, researchers will conduct within-clinic comparisons (pre- vs. post-implementation) and examine a composite of patient-level outcomes post-implementation, including the proportion of patients having any of the following 6 outcomes:
  1. receipt of a naloxone order or prescription fill;
  2. absence of opioid overdose diagnoses and naloxone administration;
  3. absence of ED visits or hospitalizations due to opioid overdose or OUD;
  4. absence of overlapping opioid and benzodiazepine use;
  5. absence of high-dose opioid use (average daily morphine milligram equivalent ≥50);
  6. receipt of referrals to non-pharmacological pain management (e.g., physical therapy, chiropractic care).
PCP's use feedback of the Overdose Prevention Alert (OPA) | From enrollment and up to 7 months post implementation of the OPA
  An online questionnaire for PCPs who interacted with OPA includes 12 Likert-scale items (4-point scale: 1 = Strongly Disagree to 4 = Strongly Agree) assessing OPA's acceptability, appropriateness, and feasibility:
  1. OPA's information was clear.
  2. OPA was easy to use.
  3. OPA helps identify patients at increased overdose risk.
  4. OPA helps understand patient's overdose risk.
  5. OPA provides risk management recommendations.
  6. OPA identifies the right patients with elevated overdose risk.
  7. OPA notifies the correct healthcare team member (i.e., PCPs).
  8. A pop-up alert is an appropriate notification approach.
  9. Signing an opioid order is the right time for OPA.
  10. Alert frequency is appropriate.
  11. I prefer OPA over the legacy naloxone alert (see picture).
  12. I want this OPA to continue to operate in my EHR.
  Mean scores (with standard deviations [SD]) will be calculated across all items, as well as individual average scores (SD).

SECONDARY OUTCOMES:
Receipt of a naloxone order or prescription fill | From enrollment and up to 12 months (3, 6, 12 months) post implementation of the Overdose Prevention Alert (OPA)
  Proportion of patients receiving alert who have a naloxone order or prescription fill
Absence of opioid overdose diagnoses and naloxone administration | From enrollment and up to 12 months (3, 6, 12 months) post implementation
  Proportion of patients receiving alert who do not have an opioid overdose diagnoses and naloxone administration
Absence of ED visits or hospitalizations due to opioid overdose or OUD | From enrollment and up to 12 months (3, 6, 12 months) post implementation
  Proportion of patients receiving alert who do not have ED visits or hospitalizations due to opioid overdose or opioid use disorder (OUD)
Absence of overlapping opioid and benzodiazepine use | From enrollment and up to 12 months (3, 6, 12 months) post implementation
  Proportion of patients receiving alert who do not have overlapping opioid and benzodiazepine use
Absence of high-dose opioid use (average daily morphine milligram equivalent ≥50) | From enrollment and up to 12 months (3, 6, 12 months) post implementation
  Proportion of patients receiving alert who do not have high-dose opioid use (average daily morphine milligram equivalent ≥50).
Receipt of referrals to non-pharmacological pain management (e.g., physical therapy, chiropractic care | From enrollment and up to 12 months (3, 6, 12 months) post implementation
  Proportion of patients receiving alert who have referrals to non-pharmacological pain management (e.g., physical therapy, chiropractic care).

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Hsuan Lo-Ciganic, PhD, Principal Investigator — Division of General Internal Medicine, School of Medicine, University of Pittsburgh, Pittsburgh, PA
Locations (1):
- University of Florida Health Internal Medicine and Family Medicine, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No
While transparency and data sharing are critical to advancing clinical research, researchers are unable to share individual participant data (IPD) derived from UF Health EHR due to institutional and legal constraints. The data are governed by strict privacy regulations, including HIPAA, which mandate the protection of patient confidentiality. Additionally, UF Health's policies restrict the dissemination of EHR data to ensure compliance with these regulations and safeguard against the risk of re-identification. As a result, while researchers can report aggregated findings, sharing raw participant-level data is not permissible under current regulatory and institutional frameworks.

REFERENCES:
- [Background] Lo-Ciganic WH, Donohue JM, Yang Q, Huang JL, Chang CY, Weiss JC, Guo J, Zhang HH, Cochran G, Gordon AJ, Malone DC, Kwoh CK, Wilson DL, Kuza CC, Gellad WF. Developing and validating a machine-learning algorithm to predict opioid overdose in Medicaid beneficiaries in two US states: a prognostic modelling study. Lancet Digit Health. 2022 Jun;4(6):e455-e465. doi: 10.1016/S2589-7500(22)00062-0. PMID 35623798
- [Background] Lo-Ciganic WH, Huang JL, Zhang HH, Weiss JC, Kwoh CK, Donohue JM, Gordon AJ, Cochran G, Malone DC, Kuza CC, Gellad WF. Using machine learning to predict risk of incident opioid use disorder among fee-for-service Medicare beneficiaries: A prognostic study. PLoS One. 2020 Jul 17;15(7):e0235981. doi: 10.1371/journal.pone.0235981. eCollection 2020. PMID 32678860
- [Background] Lo-Ciganic WH, Huang JL, Zhang HH, Weiss JC, Wu Y, Kwoh CK, Donohue JM, Cochran G, Gordon AJ, Malone DC, Kuza CC, Gellad WF. Evaluation of Machine-Learning Algorithms for Predicting Opioid Overdose Risk Among Medicare Beneficiaries With Opioid Prescriptions. JAMA Netw Open. 2019 Mar 1;2(3):e190968. doi: 10.1001/jamanetworkopen.2019.0968. PMID 30901048
- [Background] Militello LG, Diiulio J, Wilson DL, Nguyen KA, Harle CA, Gellad W, Lo-Ciganic WH. Using human factors methods to mitigate bias in artificial intelligence-based clinical decision support. J Am Med Inform Assoc. 2025 Feb 1;32(2):398-403. doi: 10.1093/jamia/ocae291. PMID 39569464
- [Background] Nguyen K, Wilson DL, Diiulio J, Hall B, Militello L, Gellad WF, Harle CA, Lewis M, Schmidt S, Rosenberg EI, Nelson D, He X, Wu Y, Bian J, Staras SAS, Gordon AJ, Cochran J, Kuza C, Yang S, Lo-Ciganic W. Design and development of a machine-learning-driven opioid overdose risk prediction tool integrated in electronic health records in primary care settings. Bioelectron Med. 2024 Oct 18;10(1):24. doi: 10.1186/s42234-024-00156-3. PMID 39420438
- See also: Center for Pharmaceutical Policy & Prescribing website — https://www.cp3.pitt.edu/